CLINICAL TRIAL: NCT03436173
Title: Investigating the Effects of the Antidepressant Fluoxetine on the Emotional Processing of Young People With Depression - a Double Blind, Placebo-controlled Design fMRI Study
Brief Title: OxSYPan: Oxford Study With Young People on Antidepressants
Acronym: OxSYPan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 12/SC/0030
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoxetine (Experimental): Fluoxetine 10 mg/2.5 ml
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Peppermint syrup measured to equivalent volume
  Interventions: Other: Peppermint syrup

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 10 mg/2.5 ml mixed with water
  Other Names: Prozac
  Arms: Fluoxetine
Other: Peppermint syrup — Liquid peppermint syrup measured to the equivalent volume and mixed with water
  Arms: Placebo

SUMMARY:
Fluoxetine is commonly used to treat adolescent depression, but the neural mechanisms underlying antidepressant drugs in the young brain are still poorly understood. This study proposes to investigate the effects of a single dose of fluoxetine on emotional neural processing in a sample of depressed adolescents, using functional Magnetic Resonance Imaging (fMRI).

DETAILED DESCRIPTION:
Depression is common in adolescence and is associated with a high risk of suicide. Clinically, the presentation of depression in young people is largely similar to the symptoms seen in adulthood, although depressed youth may exhibit increased irritability rather than (or in addition to) low mood. Therefore, irritability is included as a cardinal symptom in the diagnosis of Major Depressive Disorder (MDD) among children and adolescents but not adults (American Psychiatric Association, 2013).

Fluoxetine is the antidepressant with the most favourable benefit:risk ratio profile to treat adolescent depression, and is the only medication approved for use to treat this disorder in the United Kingdom (UK). In the United States (US), fluoxetine is also the drug of choice, together with escitalopram. However, our current understanding of the mechanisms underlying antidepressant action in adolescents and young people is poor, despite the pressing need to explain the complex patterns of clinical response to pharmacotherapy in this group.

In this randomised, placebo-controlled experimental medicine study, the investigators propose to use fMRI to investigate the early effects of fluoxetine in a sample of depressed adolescents who have been prescribed fluoxetine by their psychiatrist for the treatment of depression. Immediately after being referred to the study team, participants will be randomised to take their first dose of either fluoxetine or placebo within the study, and 6 hours later, they will undergo a neuroimaging scan.

Previous research from our group showed that a single dose of fluoxetine reduced the accuracy to detect angry facial expressions in a group of young healthy volunteers, aged 18 to 21 (Capitão et al., 2015). Given the key role of anger in the clinical presentation of adolescent depression, the reduction in anger perception following fluoxetine highlights a potential mechanism through which this antidepressant drug may exert its clinical action. However, this hypothesis remains to be investigated in depressed adolescents.

This study therefore proposes to investigate the acute effects of fluoxetine vs. placebo on emotional neural processing, specifically in response to angry faces, in a sample of adolescents with MDD. A secondary aim is to investigate the effects of fluoxetine on emotional regulation, as well as on resting-state functional connectivity.

To the extent of the investigators' knowledge, this is the first study to explore the acute neural effects of fluoxetine in depressed adolescents. This design is thought to be of high value as patients will be referred to the study immediately after being prescribed fluoxetine, therefore allowing the investigators to scan them on the day that they take their first dose of 10 mg fluoxetine or placebo, administered within the study. Patients will then start their antidepressant treatment as prescribed and managed by their treating psychiatrist. This unique time window for testing allows the investigation of the effects of fluoxetine using a placebo control, and without the ethical concerns associated with long-term antidepressant drug studies. This single dose design also enables the characterisation of the effects of fluoxetine at a time where changes in mood are not yet apparent. Indeed, the few neuroimaging studies conducted to date with depressed adolescents are limited by the absence of a placebo control and the measurement of neural changes after relatively prolonged treatments (8 weeks). Concurrent changes in symptoms make it difficult to determine whether fluoxetine has a direct effect on relevant neural regions or whether the antidepressant-induced changes in activity are an indirect consequence of mood improvement. The current study design overcomes these constraints.

The knowledge attained from this study will hopefully help increase our understanding of the early mechanisms underlying fluoxetine use in depressed adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Current episode of depression with or without comorbid anxiety and in need of antidepressant medication (as assessed by the Adolescent Psychiatrist);
* Participant and parent/legal guardian (for participants younger than 16) are willing and able to give informed consent for participation in the study;
* Male or female, aged 13-18;
* Sufficiently fluent in English to understand the task and instructions.

Exclusion Criteria:

* Current or past psychosis or mania;
* Current substance misuse;
* Psychotropic medication usage within the past 6 weeks;
* Contraindication to fMRI (e.g. metal in body, claustrophobia, pregnancy, etc);
* Risk of waiting 5-7 days before the initiation of medication assessed as posing serious risk (as assessed by the Adolescent Psychiatrist).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05-23 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2015-11-10 (Actual)

PRIMARY OUTCOMES:
Neural activity (BOLD response) in response to angry faces | 6 hours post-intervention
  fMRI data collected during a faces task involving angry, happy and fearful faces

SECONDARY OUTCOMES:
Neural activity (BOLD response) in task measuring emotional regulation | 6 hours post-intervention
  fMRI data collected during an emotional regulation task
Resting-state functional connectivity | 6 hours post-intervention
  fMRI data collected during resting-state scan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Capitao LP, Murphy SE, Browning M, Cowen PJ, Harmer CJ. Acute fluoxetine modulates emotional processing in young adult volunteers. Psychol Med. 2015 Aug;45(11):2295-308. doi: 10.1017/S0033291715000240. Epub 2015 Apr 13. PMID 25864939
- [Background] American Psychiatric Association (2013). Diagnostic and Statistical Manual of Mental Disorders, 5th edn: DSM-5. American Psychiatric Association: Arlington, VA.
- [Derived] Capitao LP, Chapman R, Filippini N, Wright L, Murphy SE, James A, Cowen PJ, Harmer CJ. Acute neural effects of fluoxetine on emotional regulation in depressed adolescents. Psychol Med. 2023 Jul;53(10):4799-4810. doi: 10.1017/S0033291722001805. Epub 2022 Jul 29. PMID 35903009